CLINICAL TRIAL: NCT03045445
Title: Comparison of Image Quality Between "Double Low-Dose" Dual Energy Liver CT and Standard Contrast Enhanced Liver CT in Patients at High-risk of HCC: Prospective, Randomized Single Center Study
Brief Title: "Double Low-Dose" DECT for HCC Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SNUH-2016-2830
Record Dates: First submitted 2017-02-04; First posted 2017-02-07 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: HCC
Keywords: CT; dual energy; low dose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Low-Dose protocol CT (Experimental): Low radiation dose + low amount of iodine contrast media at spectral CT (Philips Healthcare)
  Interventions: Diagnostic Test: Double Low-Dose protocol CT
- Standard protocol CT (Active Comparator): Standard protocol quadriphasic liver CT according to current liver CT protocol in our institution, at spectral CT (Philips Healthcare)
  Interventions: Diagnostic Test: Standard protocol CT

INTERVENTIONS:
Diagnostic Test: Double Low-Dose protocol CT — Double low-dose protocol CT (Low radiation dose quadriphasic liver CT and low dose of iodine contrast media) at spectral dual energy CT scanner
  Arms: Double Low-Dose protocol CT
Diagnostic Test: Standard protocol CT — standard protocol CT (standard dose quadriphasic liver CT and standard dose of iodine contrast media) at spectral dual energy CT scanner
  Arms: Standard protocol CT

SUMMARY:
Hypothesis: double low-dose protocol provide better lesion conspicuity than standard protocol CT in patients at high-risk of HCC.

patients who are scheduled for CECT for HCC diagnosis or surveillance are eligible for this study and allocated to either standard protocol or double-low dose protocol using spectral CT with low radiation dose and low dose of contrast media, within clinically accpetable range.

ELIGIBILITY:
Inclusion Criteria:

* high risk of HCC (chronic hepatitis B or C, or LC of any cause)
* signed informed consent
* scheduled for contrast enhanced liver CT for HCC surveillance or diagnosis

Exclusion Criteria:

* no risk factor for HCC
* history of iodine hypersensitivity
* renal dysfunction (Estimated GFR < 30mL/min/1.73m2) or on dialysis
* metformin medication within 48 hours
* any other contraindication of CE-CT
* BMI > or = 30

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Lesion conspicuity | 12 months after CT
  qualitative conspicuity assessment of focal liver lesion

SECONDARY OUTCOMES:
image noise | 12 months after CT
  qualitative analysis
beam hardening artifact | 12 months after CT
  qualitative analysis
hepatic artery conspicuity | 12 months after CT
  qualitative analysis
portal vein conspicuity | 12 months after CT
  qualitative analysis
image texture (plasticity) | 12 months after CT
  qualitative analysis
overall image quality | 12 months after CT
  qualitative analysis
presence of hepatic artery anatomic variation | 12 months after CT
  yes, no, indeterminate and if yes) describe the variation
sensitivity to detect HCC | 18 months after CT
  according to LI-RADS
radiation dose | 1 month after CT
  CTDIvol, DLP, and effective dose

OTHER OUTCOMES:
contrast media iodine amount | 1 month after CT
  contrast media iodine amount
adverse effect | 1 month after CT
  any adverse effect related with contrast media
Enhancement degree | 12 months after CT
  HU in aorta, portal vein and liver parenchyma on each phase of CT

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon JH, Chang W, Lee ES, Lee SM, Lee JM. Double Low-Dose Dual-Energy Liver CT in Patients at High-Risk of HCC: A Prospective, Randomized, Single-Center Study. Invest Radiol. 2020 Jun;55(6):340-348. doi: 10.1097/RLI.0000000000000643. PMID 31917765